CLINICAL TRIAL: NCT00682032
Title: Beta-glucan's Immuno-modulatory Effect on Non-Small Cell Lung Cancer
Brief Title: The Effect of Beta-glucan in Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Phuong T Ngo, Assistant Professor, M.D., University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08.0041; BCC-LUN-07-005 (Other: James Graham Brown Cancer Center Clinical Trials Office)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — beta-Glucans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AIM 2: subjects with suspected or definitive NSCLC diagnosis (Experimental): 1 (one) 250mg beta-glucan capsule 3 times a day for 14 days
  Interventions: Dietary Supplement: beta-glucan
- AIM 3: subjects with resectable NSCLC (Experimental): 1 (one) 250mg beta-glucan capsule 3 times a day for 10 to 20 days
  Interventions: Dietary Supplement: beta-glucan

INTERVENTIONS:
Dietary Supplement: beta-glucan — AIM 2: regimen to begin after baseline blood draw; AIM 3: regimen to begin after baseline blood draw and to be completed prior to surgery
  Other Names: Imucell WGP

SUMMARY:
The purpose of this study is to determine how beta-glucan affects the immune system in subjects with non-small cell lung cancer.

DETAILED DESCRIPTION:
Beta-glucan (Imucell WGP) is an over-the-counter dietary supplement that enhances the body's immune system. Imucell WGP is extracted from food-grade baker's yeast, which is permitted for use in food by the U.S. Food and Drug Administration (FDA). Studies in animals have shown that Imucell WGP helps trigger white blood cells to destroy cancer cells. Other animal studies combining Imucell WGP with anti-cancer medications have shown greater tumor regression and tumor-free survival.

ELIGIBILITY:
AIM 2:

Inclusion Criteria:

* suspected or definitive diagnosis of non-small cell lung cancer (NSCLC)
* treatment naive or no treatment within 6 months prior to enrollment
* able to swallow pills
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3
* absolute neutrophil count (ANC) at least 1500/microl
* able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* history of hypersensitivity reactions attributed to beta-glucan
* currently receiving continuous corticosteroids or other ongoing immunosuppressive therapy
* presence of an uncontrolled intercurrent illness including but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

AIM 3:

Inclusion Criteria:

* resectable non-small cell lung cancer (NSCLC), as determined by a thoracic surgeon
* treatment naive
* able to swallow pills
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* must be an operative candidate
* absolute neutrophil count (ANC) at least 1500/microl
* able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* history of hypersensitivity reactions attributed to beta-glucan
* currently receiving continuous corticosteroids or other ongoing immunosuppressive therapy
* presence of an uncontrolled intercurrent illness including but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-10; Primary Completion 2025-04 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
blood specimens will be obtained to examine the ability of beta-glucan to prime neutrophils complement receptor 3 (CR3) and test the cytotoxicity of the primed neutrophils. | pre-treatment and post-treatment
  compare CR3 CBRM1/5 expression, CR3-dependent cellular cytotoxicity, myeloid-derived suppressor cells (MDSC) frequency, and T-cell function (cytokine secretion) before and after beta-glucan uptake
resected lung tissue will be tested to determine macrophage phenotype | post-treatment
  AIM 3 only

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States